CLINICAL TRIAL: NCT04697693
Title: Antidepressant Response in Older Adults With Comorbid PTSD and MDD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit participants in a timely fashion due to COVID pandemic
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8111
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2022-03-28 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Post Traumatic Stress Disorder; Major Depressive Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major | interventions — Escitalopram; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with escitalopram or duloxetine (Experimental): Participant will be begun on either escitalopram 10mg or duloxetine 30mg. The default medication will be escitalopram. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the Hamilton Rating Score for Depression (HRSD) >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study. Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg of duloxetine for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study
  Interventions: Drug: Escitalopram; Drug: Duloxetine

INTERVENTIONS:
Drug: Escitalopram — The participant will be begun on either escitalopram 10mg or duloxetine 30mg. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the HRSD >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study.
  Other Names: lexapro
Drug: Duloxetine — Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study.
  Other Names: cymbalta

SUMMARY:
In the Investigator's ongoing studies of Posttraumatic Stress Disorder (PTSD) in older adults, it has been found that older adults with PTSD frequently meet the criteria for comorbid Major Depressive Disorder (MDD). Moreover, relative to trauma-exposed healthy controls (TEHCs), elders with PTSD manifest executive function deficits, fatigability, and mobility and physical function deficits that are consistent with what the investigator has observed in depressed older adults. Yet, the investigator has found that very few older adults with combined PTSD/MDD have received appropriate antidepressant treatment for their condition. These findings give rise to the questions of (1) how effective is antidepressant treatment for depressive symptoms in the context of PTSD/MDD and (2) are cognitive and physical function deficits in PTSD/MDD patients reversible with effective antidepressant treatment?

DETAILED DESCRIPTION:
Chronic PTSD in older adults leads to increased risk of mortality from cardiovascular disease, metabolic syndrome, diabetes mellitus, and ulcerative gastrointestinal disease. PTSD appears to promote aging-associated syndromes such as frailty, and older patients with PTSD exhibit faster cognitive decline and have twice the risk of dementia compared to individuals without PTSD. In addition, laboratory studies report accelerated biological signatures of aging in PTSD patients, including shortened leukocyte telomere length, increases in pro-inflammatory cytokines, and increased oxidative stress. PTSD is associated with similar anatomical brain changes to those occurring with cognitive aging, including bilateral hippocampal volume reductions, specifically affecting the dentate gyrus (DG) and CA3 subregion, and increased microvascular lesions (white matter hyperintensities [WMH]). These observations suggest that the adverse health and functional outcomes associated with chronic PTSD in older patients may be explained by a deleterious interaction between pathophysiologic changes underlying PTSD and the biology of aging, the end result of which is to accelerate senescence throughout the body and particularly in the brain. However, no prior study has explicitly tested this hypothesis by examining indices of aging in older adults with and without PTSD. In our ongoing IRB #7489, The investigator hypothesize that chronic PTSD, over and above other contributing factors, accelerates biological aging in the brain and body, leading to adverse behavioral consequences such as frailty and cognitive decline. To test these hypotheses, 150 individuals are being recruited who are aged≥50and diagnosed with PTSD. A control group of 150 age-, sex-, and trauma exposure-matched subjects without PTSD are being recruited and assessed. Included subjects undergo comprehensive neuropsychological assessment and cerebral blood volume functional magnetic resonance imaging (CBV-fMRI) to assess regional hippocampal metabolic activity and function. Structural MRI is performed to quantify WMH, regional brain volume, and cortical thickness while resting-state fMRI measures functional connectivity within hippocampal networks. PTSD subjects and controls are compared on measures of aging within the following domains: neural (DG CBV, WMH, morphology), cognitive (processing speed, memory, executive function, pattern separation), somatic (peripheral inflammatory markers, leukocyte telomere length, and measures of oxidative stress), and behavioral (grip strength, gait speed, fatigue levels). By elucidating the interaction of chronic PTSD with aging processes, data from this project may contribute to the development of rationally designed, personalized, and age-appropriate novel treatments.

Interim analyses of PTSD subjects in this study demonstrate a high degree of comorbidity with MDD. Among participants with PTSD enrolled to date, 67.1% meet the criteria for MDD and the mean Hamilton Rating Scale for Depression (HRSD) is 18.1. The most prominent cognitive differences observed to date in our study between PTSD and TEHC subjects is executive dysfunction, which is common in late-life depression.

PTSD subjects have dramatically increased fatigability and prevalence of frailty criteria compared to TEHCs, abnormalities which are also frequently seen in our older MDD samples. Yet, the investigator has found that less than 25% of these individuals are currently receiving an adequate dose and duration of first-line pharmacotherapy for MDD, while only one-third report any past medication treatment. These data raise the question of whether patients with combined PTSD/MDD could benefit from adequate antidepressant medication treatment and to what degree their cognitive and physical function deficits would be reversible with this therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Individual has completed IRB 7489
2. Diagnosed with DSM 5 MDD
3. HRSD >=18
4. Willing to and capable of providing informed consent and complying with study procedures.

Exclusion Criteria:

1. History of allergic or adverse reaction to
2. Non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20mg) and duloxetine (at least 4 weeks at dose of 60mg)during the current episode.
3. Current treatment with psychotherapy, antidepressants, or other psychotropic medications.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret R Rutherford, MD, Principal Investigator — New York State Psychiatric Institue
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With Escitalopram or Duloxetine: Participant will be begun on either escitalopram 10mg or duloxetine 30mg. The default medication will be escitalopram. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the Hamilton Rating Score for Depression (HRSD) >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study. Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg of duloxetine for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study.
  Escitalopram: The participant will be begun on either escitalopram 10mg or duloxetine 30mg. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the HRSD >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study.
  Duloxetine: Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg of duloxetine for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study.
Period: Overall Study
Arm/Group | Treatment With Escitalopram or Duloxetine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Escitalopram or Duloxetine: Participant will be begun on either escitalopram 10mg or duloxetine 30mg. The default medication will be escitalopram. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the Hamilton Rating Score for Depression (HRSD) >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study. Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg of duloxetine for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study.
  Escitalopram: he participant will be begun on either escitalopram 10mg or duloxetine 30mg. Subjects will begin escitalopram 10mg, continue this dosage for 4 weeks, then if the HRSD >7 at Week 4, he/she will have their dosage increased to 20mg for the remainder of the 8 week study.
  Duloxetine: Participants who have not responded to or not tolerated escitalopram in the current depressive episode will be started on duloxetine. They will take 30mg of duloxetine for the first 2 weeks, then, contingent on clinical assessment that the 30mg dose is sufficiently well tolerated, be increased to 60mg for the remaining 6 weeks of the study.
Arm/Group | Treatment With Escitalopram or Duloxetine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Data are not available to be reported due to patient privacy concerns.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Hamilton Rating Score for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — Scale for depressive symptoms administered by trained rater. The Hamilton is the standard measure of depression severity for clinical trials of antidepressants and was chosen to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. The scoring is based on the first 24 items of the Hamilton.
  Sum of the scores of the first 24 items (range from 0 to 74):
  0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
  units on a scale | 23 (NA) — Total number of enrolled participants is one, so standard deviation cannot be calculated.

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Score for Depression (HRSD) From Baseline to Week 8
Description: Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluating recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score above 16 is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity. The change in Hamilton Rating Score for Depression (HRSD) from baseline to week 8 was calculated as Week 8 HRSD - Baseline HRSD.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Escitalopram or Duloxetine
Number analyzed (Participants) | 1
score on a scale | 3 (NA) — Total number of enrolled participants is one, so standard deviation cannot be calculated.

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the period of 8 weeks.
Description: Subjects will have telephone/video-conference visits via a telephone and/or a HIPAA compliant video conferencing platform, Webex with the research assistant and study clinician every two weeks. If the participant requests or significant clinical worsening in the judgement of the study clinician occurs, then the participant will be brought to NYSPI for in person evaluation.
Arm/Group | Treatment With Escitalopram or Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study had a planned accrual of 25 participants but only accrued 1 participant due to challenges in recruiting during the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT04697693/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT04697693/SAP_001.pdf